CLINICAL TRIAL: NCT04659057
Title: Effect of Nebulized Lidocaine, Dexmedetomedine and Their Combination on Haemodynamics During Direct Laryngoscopy Surgery. A Randomized Controlled Clinical Trial.
Brief Title: Nebulized Lidocaine, Dexmedetomedine and Their Combination in Direct Laryngoscopy Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hala Salah El-Din El-Ozairy, MD, Lecturer of Anaesthesia, ICU and Pain management, Faculty of Medicine, Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU R 110/2020
Record Dates: First submitted 2020-11-23; First posted 2020-12-09 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Hemodynamic Instability
MeSH Terms: interventions — Dexmedetomidine; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group L (Active Comparator): Lidocaine group; 45 randomly assigned patients.
  Interventions: Drug: Nebulized Lidocaine
- Group D (Active Comparator): Demedetomidine group; 45 randomly assigned patients.
  Interventions: Drug: Nebulized dexmedetomidine
- Group DL (Active Comparator): Combined lidocaine and dexmedetomidine group. 45 randomly assigned patients.
  Interventions: Drug: Nebulized lidocaine and dexmedetomidine
- Group C (Placebo Comparator): Control group; 45 randomly assigned patients.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nebulized Lidocaine — will receive nebulized lidocaine 2%, 1 mg/kg with a maximum dose of 100 mg (5 ml).
  Other Names: Lidocaine group
  Arms: Group L
Drug: Nebulized dexmedetomidine — will receive nebulized dexmedetomidine (1 μg/kg diluted in 5 ml of saline 0.9%).
  Other Names: Dexmedetomidine group
  Arms: Group D
Drug: Nebulized lidocaine and dexmedetomidine — will receive nebulized lidocaine 2% (0.5 mg/kg) and dexmedetomidine 0.5 μg/kg dexmedetomidine in 5 ml of saline 0.9%.
  Other Names: Combined lidocaine and dexmedetomidine group
  Arms: Group DL
Other: Placebo — will receive nebulized saline 0.9% (5 ml) as control group.
  Other Names: Control group
  Arms: Group C

SUMMARY:
Direct laryngoscopy (DL) procedure is typically done under general anaesthesia as a day case. It is a short but irritating.Various drugs and drug combinations have been used to attenuate stress response to DL.Administrating nebulized form of drugs can be effective with less systemic side effects. The primary outcome of this study is to compare the effect of premedication with nebulized lidocaine, dexmedetomidine, combination of both to placebo on haemodynamic response during DL procedures.

DETAILED DESCRIPTION:
Patients will be transferred to the induction room 30 min prior to surgery. Standard monitors will be applied [pulse oximetry, non invasive blood pressure (NIBP) and electrocardiogram (ECG)]. Basal HR, systolic (SBP), diastolic (DBP) and mean arterial blood pressure (MAP) will be recorded. An intravenous 22-G cannula will be inserted, and all patients will be pre-medicated with intravenous midazolam 0.02 mg/kg, granisetrone 2mg and ranitidine 30 mg.

Patients will then be randomly and evenly allocated to one of 4 groups (45 patients each).

Nebulized solutions will be prepared by a pharmacist not participating in the study. Nebulization will be done with 100% oxygen (10 L/min) through facemask attached to a nebulizer. Patients will be asked to breath normally. Nebulization will continue till the solution in the nebulizer is all aerosolized.

Upon arrival to the operating room, routine monitors will be applied in addition to neuromuscular monitor and end tidal CO2 (ETCO2). General anaesthesia will be induced, after 5 min of preoxygenation, by intravenous fentanyl 1 μg/kg, propofol 1.5-2 mg/kg titrated to a loss of verbal response and rocuronium 1 mg/kg to facilitate endotracheal intubation. Mackintosh laryngoscope will be introduced when train of four (TOF) count reaches 1. High volume-low pressure endotracheal tube (size 5-5.5) will be inserted by senior anaesthesiologist. HR, SBP, DBP and MAP will be recorded immediately after intubation.

Anaesthesia will be maintained by sevoflurane 2-3% in oxygen to air ratio 1:1. Rocuronium 0.1 mg/kg when required. Positive pressure ventilation will be set to maintain ETCO2 30-35 mmHg.

SBP, DBP, MAP and HR will be recorded on arrival to the induction room (baseline), after endotracheal intubation, and then every 5 min throughout the surgery.

In case of hypertension (defined as SBP > 140 mmHg, DBP >90 mmHg or MAP 20% higher than baseline) and/or tachycardia (defined as HR 20% higher than baseline), boluses fentanyl 0.5 μg/kg will be given with a maximum dose of 2 μg/Kg. If hypertension and/or tachycardia continue after reaching the maximum dose of fentanyl, loading dose of esmolol 500 μg/Kg will be started, followed by infusion of 100-300 μg/kg/min. The use and total dose of esmolol will be recorded.

In cases of significant hypotension (defined as mean blood pressure < 70 mmHg), the patient will be treated initially with an intravenous (IV) fluid bolus of10 mL/kg normal saline, and if the condition persists, the patient will given 0.1-0.3 mg/kg IV ephedrine, which will be repeated every 3-5 minutes until the blood pressure is normalized. Significant bradycardia (defined as heart rate < 60 beat/min) will be treated, when needed, with IV atropine 0.02 mg/kg.

At the conclusion of surgery, sevoflurane will be discontinued and patients will inhale 100% O2. After return of spontaneous breathing, residual neuromuscular block will be reversed with intravenous neostigmine 0.05 mg/kg and glycopyrolate 0.01 mg/kg. Extubation will be done when the patient starts to show purposeful movements.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients admitted for DL surgery.

Exclusion Criteria:

* Uncontrolled hypertension (MAP > 100 mmHg) or ischaemic heart disease.
* End stage renal impairment.
* Chronic drug or alcohol abuse.
* Predicted difficult airway, laryngoscopy and intubation time > 30 sec, more than one attempt of intubation.
* Morbid obesity (BMI > 30).
* Known allergy to the drugs used.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-07-11 (Actual); Study Completion 2021-07-11 (Actual)

PRIMARY OUTCOMES:
Heart Rate | Every 5 minutes for 30-60minutes
  Heart rate in beats/min
Systolic blood pressure | Every 5 minutes for 30-60 minutes
  Systolic blood pressure in mmHg
Diastolic blood pressure | Every 5 minutes for 30-60 minutes
  Diastolic blood pressure in mmHg
Mean arterial pressure | Every 5 min for 30-60 minutes
  Mean arterial pressure in mmHg

SECONDARY OUTCOMES:
Total fentanyl and esmolol consumption | For 30-60 minutes
  The total dose of fentanyl and/or esmolol consumed by each patient
recovery time | 5- 15 minutes
  The time from discontinuation of anaesthetic drugs until response to verbal commands

CONTACTS AND LOCATIONS:
Overall Officials: Hala S El-Ozairy, MD, Principal Investigator — Ain Shams University
Locations (2):
- Egypt (2):
  - Ain Shams University, Cairo, Cairo Governorate
  - Ain Shams University Hospitals, Cairo